CLINICAL TRIAL: NCT02191787
Title: Pharmacokinetic-pharmacodynamic Assessment of Seresis® o.d.: an Open, Uncontrolled, Non-randomised Intraindividual Pilot-study
Brief Title: Pharmacokinetic-pharmacodynamic Assessment of Seresis® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1135.2
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (1):
- Seresis® + Placebo (Experimental): 2 capsules Seresis® o.d. for 5 days
  2 capsules Placebo o.d. the day before treatment with Seresis®
  Interventions: Drug: Seresis®; Drug: Placebo

INTERVENTIONS:
Drug: Seresis®
Drug: Placebo

SUMMARY:
Study to determine the antioxidant potency of Seresis® in the serum of healthy volunteers and the optimal time for blood sampling

ELIGIBILITY:
Inclusion Criteria:

The subjects to be enrolled are healthy volunteers, defined as follows:

* Healthy men or women between 18 and 30 years old
* Non-smokers
* Fit for work
* Having given informed consent and signed the form

Exclusion Criteria:

* Any serious disorder that might interfere with his/her participation in this study and the evaluation of the safety of the test drug (e.g. renal insufficiency, hepatic dysfunction, cardiovascular disease, hypervitaminosis A, psychic disorder etc.).
* Treatment with other drug that might interfere with the evaluation of the safety of the test drug
* Known hypersensitivity to any of the ingredients of the study drug
* Pregnancy, lactation, women of childbearing potential who do not use an established contraceptive
* Drug and alcohol abuse
* Participation in another trial
* Known abnormal values of the laboratory tests (if detected after enrolment, subjects will continue the treatment provided there are not medical objections)
* Specific dietary requirements that do not allow the volunteers to meet the dietary guidelines set out for this study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1998-03; Primary Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Changes in total antioxidant activity of Seresis® | Baseline, Day 2
  determined by chemoluminescence

SECONDARY OUTCOMES:
Changes in total antioxidant activity of Seresis® | Day 2, day 6
  determined by chemoluminescence
Assessment of tolerability on a 4-point scale | Day 14
Number of patients with abnormal changes in laboratory parameters | up to day 14
Number of patients with adverse events | up to day 14